CLINICAL TRIAL: NCT07019168
Title: The Effects of Blood Flow Restriction-Based Jump Squat Exercise on Performance Parameters in Elite Volleyball Players: A Prospective Randomized Controlled Trial
Brief Title: The Effects of the Blood Flow Restriction Method on Performance Parameters in Elite Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Süreyyapaşa Sports Club (Unknown)
Responsible Party: Principal Investigator, Furkan ÖZKUL, Master's Student in Physiotherapy, Bahçeşehir University, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BAU-FTR-FO-01
Record Dates: First submitted 2025-06-03; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Jump Performance, Agility, Balance, Blood Flow Restriction, Fatigue
Keywords: Jump Squat; Blood Flow Restriction; BFR; Agility; Balance; Vertical Jump; Fatigue; Plyometric Training; Volleyball; Performance
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two parallel groups: one group performed jump squat exercises with blood flow restriction (BFR), and the other group performed the same exercises without BFR. Both groups followed the same protocol over a 4-week period.
Masking Description: No masking was applied in this study. All participants and investigators were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants performed the same jump squat protocol without blood flow restriction. Training frequency and duration matched the BFR group.
  Interventions: Behavioral: Jump Squat without Blood Flow Restriction
- BFR Group (Experimental): Participants in this group performed jump squat exercises with blood flow restriction (BFR) using a manually adjustable, non-automated tourniquet placed on the proximal region of both thighs. The training protocol consisted of 3 sets of 10 repetitions, carried out 3 times per week for 4 weeks. Each session was preceded by a standardized warm-up routine including dynamic stretching and general activation exercises. The BFR was applied during the exercise to partially restrict venous return while maintaining arterial inflow, creating a hypoxic environment in the working muscles.
  Interventions: Behavioral: Jump Squat with Blood Flow Restriction (BFR)

INTERVENTIONS:
Behavioral: Jump Squat with Blood Flow Restriction (BFR) — This intervention consisted of jump squat exercises performed with blood flow restriction applied using a non-automated, manually adjustable tourniquet placed on the proximal thighs. The restriction was applied during the exercise to partially limit venous return while maintaining arterial flow. The exercise protocol included 3 sets of 10 repetitions, performed 3 times per week for 4 weeks. A standardized warm-up preceded each session.
  Other Names: BFR Training
  Arms: BFR Group
Behavioral: Jump Squat without Blood Flow Restriction — This intervention consisted of the same jump squat protocol as the experimental group but without the application of blood flow restriction. Participants performed 3 sets of 10 repetitions, 3 times per week for 4 weeks. Each session was preceded by a standardized warm-up routine that included dynamic stretching and general activation exercises.
  Other Names: Classic Jump Squat
  Arms: Control Group

SUMMARY:
This study aims to investigate the effects of blood flow restriction (BFR) applied during jump squat exercises on selected performance parameters in elite volleyball players. Prior to each training session, all participants followed a standardized warm-up protocol that included dynamic stretching, mobility exercises, and general body activation to prepare for the workout. Following this preparation phase, the jump squat exercises were performed.

Participants were randomly assigned to two groups. The experimental group performed the jump squats under blood flow restriction using a manually controlled, non-automated tourniquet, while the control group performed the same exercises without any restriction.

Performance parameters were assessed before and after the 4-week intervention using the following measurement tools:

Jump performance: Measured using the Optojump system

Agility: Assessed with the Hexagon Agility Test

Balance: Evaluated using the Y Balance Test

Perceived fatigue: Measured via the Borg Rating of Perceived Exertion (RPE) scale

The purpose of the study is to determine whether jump squat exercises performed under BFR conditions can lead to greater improvements in athletic performance and perceived fatigue compared to traditional training methods. The study was conducted using equipment provided by Bahçeşehir University and included licensed volleyball players from Süreyyapaşa Sports Club. The research protocol was approved by the Non-Interventional Research Ethics Committee of Üsküdar University.

DETAILED DESCRIPTION:
This study aims to investigate the effects of jump squat exercises performed with the blood flow restriction (BFR) method on jump performance, agility, balance, and perceived fatigue in volleyball players. The effectiveness of the BFR method on these performance parameters was evaluated in comparison to classical training methods.

The study was conducted on 22 male volleyball players actively training at Süreyyapaşa Sports Club, who had similar age and training backgrounds. Participants were randomly assigned into two equal groups of 11: the experimental group (BFR group), which performed jump squats with blood flow restriction, and the control group, which performed the same exercises without restriction.

All participants followed the same exercise protocol for four weeks, training three times per week. Before each training session, a standardized warm-up routine including dynamic stretching, mobility, and general activation exercises was applied. Following the warm-up, participants performed jump squat exercises in 3 sets of 10 repetitions. In the BFR group, a manually adjustable, non-automated tourniquet device was applied to the proximal region of both thighs during the exercise. This partially maintained arterial flow while restricting venous return, thereby creating a hypoxic environment in the target muscles. No tourniquet was used in the control group.

Pre- and post-intervention assessments were performed using the following measurement tools:

Jump performance was measured using the Optojump system to assess vertical jump height.

Agility was assessed with the Hexagon Agility Test.

Balance was evaluated using the Y Balance Test, targeting lower extremity stability.

Perceived fatigue was recorded using the Borg Rating of Perceived Exertion (RPE) scale.

The aim of this study was to comparatively evaluate the performance outcomes of jump squat exercises with and without BFR in trained volleyball players. Data were statistically analyzed to determine whether the inclusion of BFR provided measurable benefits in terms of explosive strength, agility, balance, and fatigue. The findings of this study are expected to contribute to the development of safer and more effective training protocols for improving athletic performance.

This research was approved by the Üsküdar University Non-Interventional Research Ethics Committee. All measurement and test devices used in the study were provided by Bahçeşehir University. The training sessions were carried out using the infrastructure of the Süreyyapaşa Sports Club.

ELIGIBILITY:
Inclusion Criteria:

* Male volleyball players aged 18 to 25
* Playing volleyball regularly for at least 3 years
* No musculoskeletal injury in the past 6 months
* Physically capable of completing the training and testing protocol
* Willing to participate and having signed the informed consent form

Exclusion Criteria:

* History of serious musculoskeletal injury or surgical intervention in the past 6 months
* Presence of chronic diseases (e.g., cardiovascular diseases, diabetes, joint disorders)
* Physical or psychological conditions that may prevent safe participation during exercise
* Inability to adhere to the exercise protocol throughout the study
* Presence of any contraindication to blood flow restriction training, including:

Smoking,History of venous thromboembolism,Risk of peripheral vascular disease (Ankle-Brachial Index < 0.9),Body mass index (BMI) ≥ 30 kg/m²

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Height | Baseline and post-intervention (after 4 weeks of training)
  Vertical jump height was measured using the Optojump Next System. The system records jump height in centimeters based on flight time. Higher values indicate better performance (higher jump). There is no fixed maximum value, as the outcome depends on individual athletic ability.

SECONDARY OUTCOMES:
Agility (Hexagon Agility Test) | Baseline and post-intervention (after 4 weeks of training)
  Agility was assessed using the Hexagon Agility Test. The total time to complete the test was recorded in seconds. Lower times indicate better performance (better outcome). There is no fixed minimum, but the theoretical minimum would approach zero; no upper limit is predefined.
Dynamic Balance (Y Balance Test) | Baseline and post-intervention (after 4 weeks of training)
  Balance was evaluated using the Y Balance Test for the lower extremity. Reach distances were measured in centimeters for each leg in anterior, posteromedial, and posterolateral directions. Higher scores indicate better balance (better outcome). There is no fixed maximum value as it depends on individual performance.
Perceived Fatigue (Borg RPE Scale) | Baseline and post-intervention (after 4 weeks of training)
  Perceived fatigue was measured using the Borg Rating of Perceived Exertion (RPE) Scale, which ranges from 6 to 20, where higher scores indicate greater perceived exertion (worse outcome). Participants reported their perceived level of exertion before and after the 4-week intervention (pre- and post-intervention measurements).

CONTACTS AND LOCATIONS:
Overall Officials: Gokay GORMELI, MD, PhD, Principal Investigator — Bahçeşehir University, Faculty of Health Sciences; Melike Gizem KALAYCI, PhD, PT, Principal Investigator — Bahçeşehir University, Faculty of Health Sciences
Locations (1):
- Süreyyapaşa Sports Club, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy considerations and because data sharing is not planned as part of this study's dissemination strategy.